CLINICAL TRIAL: NCT00100919
Title: Coupled Joint Proprioception and Multi-Joint Movement in the Lower Extremity: A Pilot Study
Brief Title: Sensing of Leg Position and Movement
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050042; 05-CC-0042
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-07-06

CONDITIONS: Proprioception
Keywords: Kinesithesia; Sensorimotor Function; Somatosensory; Muscle Spindles; Sensory Feedback; Healthy Volunteer; HV

SUMMARY:
This study will collect information on how people sense leg position and movement. The findings may help scientists develop better ways to evaluate and treat joint problems.

Healthy adult volunteers between 21 and 40 years of age may be eligible for the study. Candidates are screened with a brief questionnaire and examination to determine their strength, flexibility, and sensation.

Participants sit on a specially designed chair, with their foot and leg placed in a custom-made apparatus that controls knee and ankle movements. The skin is marked to indicate the area of interest for ultrasound assessment of muscle. Subjects respond to joint position changes for several trials. The procedure takes a maximum of 2.5 hours to complete.

...

DETAILED DESCRIPTION:
Proprioception can be described as afferent information typically arising from peripheral mechanoreceptors that contribute to postural control, joint stability and conscious sensation of movement. Sensation of movement can be further divided into joint position sense (JPS) and the detection of passive movement sense (DPMS). Collectively, these two sensory modalities are commonly referred to as joint kinesthesia. Joint kinesthesia appears dependent on specific joint anatomical structure, suggesting different levels of acuity among various joints. However, whole limb accuracy appears to be greater than summed error across multiple joints of an extremity. Some suggest that it is only JPS errors greater than 3 degrees that have any functional significance on gait. However, the authors' calculations of position error on gait neglect JPS errors from the ankle and hip, which could also severely influence whole limb position sense, impacting gait. We believe that the central nervous system (CNS) links together afferent proprioceptive feedback from multiple joints of a limb segment to reduce kinesthetic error across a whole limb. The redundancy of the afferent information can be used as an "error check" to improve proprioceptive feedback in order to maintain function. We have used the term Coupled Joint Proprioception (CJP) in order to describe this phenomenon.

To better understand the relationship between CJP and human function, we would have to isolate movement at two adjacent joints, while controlling bi-articular muscle length, to determine its influence on single joint kinesthesia. Bi-articular muscles provide a mechanical linkage within a limb to transfer forces. Afferent information from bi-articular muscles in particular could provide a context with which proprioceptive information from other structures (single joint muscles, joint or cutaneous receptors) can maintain or enhance proprioception within a limb. The redundant information, provided by the two-joint muscles, is the basis on which we describe CJP.

The overall objective of this non-invasive pilot study is to establish the methodology necessary to test the influence of CJP on knee joint kinesthesia and proprioceptive capabilities. The primary goal is to establish two experimental conditions in which similar motions of simultaneous knee joint extension and ankle joint plantar flexion result in shortening and lengthening of all gastrocnemius muscle fibers. Following establishment of these conditions, the second goal is to develop and evaluate novel methods for studying the influence of CJP on the detection of passive movement and joint position sense at the knee joint. The information from this pilot data will also help determine the total number of subjects required to undertake a larger clinical investigation of the CJP phenomenon.

It is important to study CJP, as proprioception is typically measured clinically at a single joint in human subjects. Human function usually incorporates multiple joints, suggesting that CJP, measured across two joints, could be more representative of human proprioceptive function. Therefore, CJP would provide an avenue to better study the influence of proprioceptive feedback on human function such as walking. This is especially important because maintaining proprioceptive feedback while walking may minimize falls in patients who are at risk due to lower extremity injuries or pathologies.

ELIGIBILITY:
* INCLUSION CRITERIA

This study will include healthy males and females between 21 and 40 years of age. This age range is scientifically justified as both the CNS and musculoskeletal system are not fully matured until adulthood while lower extremity proprioception is reported to decrease with older subjects. For this project the term healthy is defined as a lack of systemic disease that alters ability of subjects to participate in activities of their choice. In addition, healthy means no current pathology where there is any possibility of damage to muscle, ligament or cartilage in the lower extremity.

EXCLUSION CRITERIA

Subjects with a history of lower extremity musculoskeletal injury, which can alter peripheral feedback from cutaneous joint or muscle mechanoreceptors, will be excluded from this study. This includes a recent history of chronic or severe lower extremity injuries such as recent surgery, trauma, degenerative joint changes, which could influence performance in this study. Examples of exclusions include ankle sprains and patella dislocations and subjects will be excluded if they have experienced these injuries within the last six months. Multiple (greater than 3) injuries, such as those described, would warrant exclusion as this could be an indicator of impaired sensation or long term deficit. The presence of local pain or the presence of an impaired sensation, indicating possible CNS dysfunction will also exclude subjects from this study. Subjects with pain will be identified the screening form while subjects with impaired sensation, indicating CNS dysfunction, will be identified by Part 2, or the physical examination of the screening form. This screening form will also evaluate general muscle strength, range of motion, sensation and the joint integrity. This pilot study will use a total of thirty subjects. Subjects will also be screened for excessive hamstring tightness, as the position described above could produce some discomfort with prolonged subject positioning.

This investigation is intended to develop methodology and obtain pilot data regarding the existence of coupled proprioception in mature healthy adults. Therefore, subjects below the age of 21 are excluded, as a developing musculoskeletal and central nervous system could impact the outcome of this study.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2005-01-04; Study Completion 2010-07-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barrack RL, Skinner HB, Brunet ME, Haddad RJ Jr. Functional performance of the knee after intraarticular anesthesia. Am J Sports Med. 1983 Jul-Aug;11(4):258-61. doi: 10.1177/036354658301100414. PMID 6614298
- [Background] Barrack RL, Skinner HB, Brunet ME, Cook SD. Joint kinesthesia in the highly trained knee. J Sports Med Phys Fitness. 1984 Mar;24(1):18-20. No abstract available. PMID 6471834
- [Background] Barrack RL, Skinner HB, Cook SD. Proprioception of the knee joint. Paradoxical effect of training. Am J Phys Med. 1984 Aug;63(4):175-81. PMID 6465302